CLINICAL TRIAL: NCT02970838
Title: Evaluation of a Structured Weight-loss Program for Therapy of Obesity and Diabetes Mellitus Type 2
Brief Title: Therapy of Obesity and Diabetes Mellitus Type 2
Acronym: TADIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BB62/12a
Record Dates: First submitted 2016-11-01; First posted 2016-11-22 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Obesity; Diabetes Type 2; Weight Loss
Keywords: Formula diet
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): Patients take part in a structured weight-loss program over 15 weeks including a fasting phase with formula diet over six weeks
  Interventions: Other: Structured weight-loss program

INTERVENTIONS:
Other: Structured weight-loss program — During the fasting phase, daily consumption consists of five sachets fully replacing normal food and corresponded to an energy content of 800 kcal. This fasting phase is followed by a four-week refeeding phase, during which regular food will be reintroduced and formula diet is gradually replaced until a daily total intake of 1200 kcal is reached. During the last five weeks of the program, energy intake is gradually increased to an individual level between 1200 kcal and 1500 kcal that allowed subjects to keep their weight stable.
  Once a week participants visit the study center to monitor health status and taking part in supervised exercises and a nutritional and behavioral counseling.
  Other Names: OPTIFAST II Short Program

SUMMARY:
To evaluate a standardized weight-loss program as treatment option for obesity and type 2 diabetes, changes in body composition and metabolic control are investigated in obese patients with diabetes.

DETAILED DESCRIPTION:
Men and women with obesity and diabetes mellitus type 2 are invited to join a standardized weight-loss program (six weeks of formula diet, followed by the reintroduction of regular food with gradually increasing energy intake over nine weeks) for a duration of 15 weeks. All subjects undergo bioelectrical impedance analyses to investigate body composition and magnet resonance imaging to measure fat mass and fat fractions of abdominal organs, at three time points: first before the program, then at the end of the six weeks of formula diet and finally, at the end of the program after 15 weeks. Laboratory data are measured before and after the program.

ELIGIBILITY:
Inclusion Criteria:

* known type 2 diabetes
* body-mass-index between 27 and 45 kg/m²

Exclusion Criteria:

* treatment with incretin mimetic drugs < 3 month
* pregnancy
* immobilization
* severe heart, liver or renal failure
* dementia
* eating disorder
* alcoholism

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-11; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c value | measured at week 0 and 15

SECONDARY OUTCOMES:
Change in weight | measured at week 0, 6 and 15
Change in body-mass-index | measured at week 0, 6 and 15
Change in waist circumference | measured at week 0, 6 and 15
Change in hip circumference | measured at week 0, 6 and 15
Change in body composition | measured at week 0, 6 and 15
  Body composition will be assessed with bioimpedance
Change in fat fractions of abdominal organs | measured at week 0, 6 and 15
  Fat fraction of abdominal organs will be assessed with magnet resonance imaging
Change in visceral fat volume | measured at week 0, 6 and 15
  Visceral fat volume will be assessed with magnet resonance imaging
Change in fasting glucose | measured at week 0 and 15
Change in fasting insulin | measured at week 0 and 15
Change in triglycerides | measured at week 0, 6 and 15
Change in cholesterol | measured at week 0, 6 and 15
Change in HDL cholesterol | measured at week 0, 6 and 15
Change in LDL cholesterol | measured at week 0, 6 and 15
Change in alanine transaminase | measured at week 0, 6 and 15
Change in aspartate transaminase | measured at week 0, 6 and 15
Change in gamma-glutamyl transferase | measured at week 0, 6 and 15
Change in alkaline phosphatase | measured at week 0, 6 and 15
Change in uric acid | measured at week 0, 6 and 15
Change in 25-hydroxy-vitamine d3 | measured at week 0 and 15
Change in 1,25-dihydroxy-vitamine d3 | measured at week 0 and 15
Change in plasma calcium | measured at week 0 and 15
Change in plasma phosphate | measured at week 0 and 15
Change in insulin-like growth factor-1 | measured at week 0 and 15
Change in testosterone | measured at week 0 and 15
Change in sex hormone-binding globulin | measured at week 0 and 15
Change in quality of life | measured at week 0 and 15
  Quality of life was determined using SF-12
Change in sleep quality | measured at week 0 and 15
  Sleep quality was determined using the Pittsburgh sleep quality index
Change in diet history | measured at week 0 and 15
  7-day food record brought in at weeks 0 and 15 will be analyzed for macronutrient intake

CONTACTS AND LOCATIONS:
Overall Officials: Markus M Lerch, MD, Principal Investigator — Department of Medicine A, University Medicine Greifswald
Locations (1):
- University Medicine Greifswald, Greifswald, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Frost F, Storck LJ, Kacprowski T, Gartner S, Ruhlemann M, Bang C, Franke A, Volker U, Aghdassi AA, Steveling A, Mayerle J, Weiss FU, Homuth G, Lerch MM. A structured weight loss program increases gut microbiota phylogenetic diversity and reduces levels of Collinsella in obese type 2 diabetics: A pilot study. PLoS One. 2019 Jul 18;14(7):e0219489. doi: 10.1371/journal.pone.0219489. eCollection 2019. PMID 31318902